CLINICAL TRIAL: NCT04976244
Title: Collaborative Ocular Antiangiogenic Study of Ukraine. Multicentral, Open-label, Randomized, Prospective Study of Antiangiogenic Therapy of Choroidal Neovascularisation Associated With Pathologic Myopia
Brief Title: Brolucizumab for CNV Associated With Pathologic Myopia
Acronym: COASTUAbaCNV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Odessa National Medical University (Other); Mykolaiv Region Ophthalmogical Hospital (Other); Central Polyclinic of Internal Affairs of Ukraine (Other Government); Lesya Ukrainka Volyn National University (Other)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, Head of Laser Department, The Filatov Institute of Eye Diseases and Tissue Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0118U001612m
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Pathologic Myopia
Keywords: fundus diseases; antiangiogenic therapy; choroidal neovascularization; pathologyc myopia; intravitreal injection; anti-VEGF; brolucizumab; aflibercept
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Intravitreal Injections; Refractometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab (Active Comparator): Arm B
  Interventions: Procedure: Intravitreal injection
- Aflibercept (Active Comparator): Arm A
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intravitreal injection — Intravitreal injection to the regimen pro re nata
  Other Names: Patients after general ophthalmic examination (visometry, refractometry, biomicroscopy, ophthalmoscopy, OCT, FA) receive injections according to the regimen pro re nata from the initial injection.

SUMMARY:
The purpose of this study is to determine the effectiveness of antiangiogenic therapy to choroidal neovascularization secondary to pathologic myopia.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of antiangiogenic therapy to choroidal neovascularization secondary to pathologic myopia.

This study is planned as a randomized, multicenter, open-label, comperative, interventional. Patients with myopia included in it will receive brolucizumab or aflibercept.

The treatment proposed in this study is based on the world experience and scientific developments of the Filatov Institute of Eye Diseases and Tissue Therapy of the NAMS of Ukraine". Therefore, it is expected that the benefit/risk ratio in relation to the participation in this study should not be different from that described in the scientific literature and the benefits outweigh the risk. It is known that the absence of treatment in these diseases leads to an irreparable loss of central vision.

Patients with a pathologic myopia with CNV (native) will be treated with antiangiogenic drugs according to the regimen pro re nata.

ELIGIBILITY:
Inclusion Criteria:

* Able to read (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent form or a family member) and understand the informed consent form and willing to sign the informed consent form.
* Signed informed consent form.
* Men and women ≥ 18 years of age.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* Myopia of greater than or equal to -6 D OR axial length of greater than (if the spherical myopic equivalent is <6.0 diopters, then the patient should have myopic changes in the macula: lacquer cracks, focal chorioretinal atrophy, posterior staphyloma) or equal to 26.5 mm.
* Active subfoveal or juxtafoveal (within 1 to 199 μm of the center of the fovea) CNV secondary to pathologic myopia as defined by leakage on FA.
* Transparent optical media and possibility to mydriasis.
* Best corrected visual acuity at least 20/200 Equivalent of Snellen (ETDRS).

Exclusion Criteria:

* Ocular media of insufficient quality to obtain fundus and OCT images in the study eye
* Recurrent mCNV in the study eye
* History or presence of CNV with an origin other than pathologic myopia in the study eye
* Ocular inflammation or external ocular inflammation in the study eye
* Concurrent disease in the study eye that would compromise BCVA or require medical or surgical intervention during the study period
* Any ocular disorder in the study eye that, in the opinion of the investigator, may confound interpretation of the study results
* Significant scarring or atrophy in the fovea that indicates substantial irreversible vision loss in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Evidence at examination of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye or current treatment for serious systemic infection
* Vitreomacular traction or traction retinal detachment, epiretinal membrane in either eye
* Any iris neovascularization and/or vitreous hemorrhage in either eye
* Uncontrolled glaucoma, or previous filtration surgery in either eye
* Prior and concomitant treatments
* Any prior or concomitant treatment with another investigational agent for mCNV in the study eye.
* Any previous panretinal photocoagulation or subfoveal thermal laser therapy in the study eye.
* Any prior treatment with photodynamic therapy in the study eye.
* Cataract surgery within 3 months prior to Day 1 in the study eye.
* Yttrium-aluminum-garnet laser capsulotomy within 2 months prior to Day 1 in the study eye.
* Any other intraocular surgery within 3 months prior to Day 1 in the study eye.
* History of vitreoretinal surgery and/or scleral buckle surgery in the study eye.
* Any prior treatment with anti-VEGF agents
* Previous use of intraocular or periocular corticosteroids in either eye within 3 months prior to Day 1
* Previous assignment to treatment during this study
* Uncontrolled hypertension
* History of cerebrovascular disease or myocardial infarction within 6 months prior to Baseline/Day 1
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect interpretation of the results of the study, or renders the subject at high risk from treatment complications
* Women of childbearing potential without contraception, women who intend to breastfeed during the study. All subjects (both men and women) of childbearing potential who are unwilling to use adequate birth control measures during the course of the study.
* Renal failure requiring dialysis or renal transplant
* Participation in an investigational study within 30 days prior to Screening/Visit 1 that involved treatment with any drug (excluding vitamins and minerals) or device
* Known serious allergy to the fluorescein sodium for injection in angiography or Verteporfin
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS Chart | Baseline-Month 12
  Defined study baseline range of ETDRS equivalent of 20/200 to 20/20) in the study eye; a higher score represents better functioning.

SECONDARY OUTCOMES:
Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) | Baseline-Month 12
  A negative number indicates improvement (reduced thickness).
Average Number of Intravitreal Injections | Baseline-Month 12
  The number of intravitreal injections administered
Number of Inflamations after Intravitreal Injections | Baseline-Month 12
  The number of inflamations registered in patients after intravitreal injections

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (4):
- Ukraine (4):
  - Lesya Ukrainka Volyn National University, Lutsk
  - Mykolaiv Region Ophthalmogical Hospital, Mykolaiv
  - Odessa National Medical University, Odesa
  - The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korol AR, Zadorozhnyy OS, Naumenko VO, Kustryn TB, Pasyechnikova NV. Intravitreal aflibercept for the treatment of choroidal neovascularization associated with pathologic myopia: a pilot study. Clin Ophthalmol. 2016 Nov 4;10:2223-2229. doi: 10.2147/OPTH.S117791. eCollection 2016. PMID 27853350